CLINICAL TRIAL: NCT00223691
Title: Evaluation and Treatment of Autonomic Failure.
Brief Title: Treatment of Orthostatic Hypotension in Autonomic Failure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor of Medicine and Pharmacology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 000814; HL46681
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Autonomic Failure; Orthostatic Hypotension
Keywords: orthostatic hypotension; autonomic failure
MeSH Terms: conditions — Pure Autonomic Failure; Hypotension, Orthostatic | interventions — Atomoxetine Hydrochloride; Acarbose; Pyridostigmine Bromide; Yohimbine; Midodrine; Modafinil; Octreotide; Drinking; Diphenhydramine; Ranitidine; Tranylcypromine; caffeine, ergotamine drug combination; Celecoxib; Pseudoephedrine; Methylphenidate; Indomethacin; Ibuprofen; Oxymetazoline; Acetazolamide; Rivastigmine; carbidopa, levodopa drug combination; Carbidopa

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: active intervention (Experimental): atomoxetine, pyridostigmine bromide, yohimbine, midodrine hcl, modafinil, octreotide, water intake, ranitidine hcl, diphenhydramine hydrochloride, tranylcypromine, ergotamine/ caffeine, celecoxib, pseudoephedrine, methylphenidate, indomethacin, ibuprofen, Oxymetazoline 0.05% nasal solution, acarbose, Rivastigmine tartrate, acetazolamide, carbidopa/levodopa, inflatable abdominal binder or bovril
  Interventions: Drug: Atomoxetine; Drug: Acarbose; Drug: Pyridostigmine Bromide; Drug: Yohimbine; Drug: Midodrine HCl; Drug: Modafinil; Drug: Octreotide; Other: water intake; Drug: Diphenhydramine Hydrochloride; Drug: Ranitidine HCL; Drug: Tranylcypromine; Drug: Ergotamine/ Caffeine; Drug: Celecoxib; Drug: Pseudoephedrine; Drug: Methylphenidate; Drug: Indomethacin; Drug: Ibuprofen; Drug: Oxymetazoline 0.05% nasal solution; Dietary Supplement: Bovril; Drug: Acetazolamide; Drug: Rivastigmine tartrate; Drug: Carbidopa/levodopa; Device: Inflatable abdominal binder
- 2: Placebo or sham device (Placebo Comparator): placebo pill or inflatable abdominal binder (sham)
  Interventions: Drug: placebo; Device: inflatable abdominal binder (sham)

INTERVENTIONS:
Drug: Atomoxetine — 10-50 mg, PO. Single dose. Alone or in combination with Yohimbine or Mestinon.
  Other Names: Strattera
  Arms: 1: active intervention
Drug: Acarbose — 25-100 mg, PO. Single dose.
  Other Names: Precose
  Arms: 1: active intervention
Drug: Pyridostigmine Bromide — 30 mg-180 mg PO. Single dose. Alone or in combination with Yohimbine or atomoxetine.
  Other Names: Mestinon
  Arms: 1: active intervention
Drug: Yohimbine — 2.7, 5.4 or 10.8 mg PO. Single dose. Alone or in combination with Atomoxetine or Pyridostigmine.
  Other Names: Yocon
  Arms: 1: active intervention
Drug: Midodrine HCl — 2.5, 5.0, 7.5, 10 mg PO. Single dose
  Other Names: ProAmatine
  Arms: 1: active intervention
Drug: placebo — PO.Single dose.
  Arms: 2: Placebo or sham device
Drug: Modafinil — 50-400 mg PO. Single dose
  Other Names: Provigil
  Arms: 1: active intervention
Drug: Octreotide — 5-50 µg, S.C. Single dose.
  Other Names: Sandostatin
  Arms: 1: active intervention
Other: water intake — Tap water 2 onz., 8 oz., 16 oz. PO, alone or in combination with any of the above medications. Single dose.
  Arms: 1: active intervention
Drug: Diphenhydramine Hydrochloride — 12.5 mg-100 mg PO. Single dose. Alone or in combination with Ranitidine
  Other Names: Benadryl
  Arms: 1: active intervention
Drug: Ranitidine HCL — 150-300 mg PO. Single dose. Alone or in combination with Diphenhydramine.
  Other Names: zantac
  Arms: 1: active intervention
Drug: Tranylcypromine — 5 - 40 mg PO. Single dose
  Other Names: Parnate
  Arms: 1: active intervention
Drug: Ergotamine/ Caffeine — Ergotamine: 1.0 mg PO. Single dose. Caffeine 100 mg PO.Single dose
  Other Names: Cafergot
  Arms: 1: active intervention
Drug: Celecoxib — 50-200 mg PO. Single dose
  Other Names: Celebrex
  Arms: 1: active intervention
Drug: Pseudoephedrine — 15, 30 or 60 mg, PO. Single dose.
  Other Names: Sudafed
  Arms: 1: active intervention
Drug: Methylphenidate — 5 or 10 mg PO. Single dose.
  Other Names: Ritalin
  Arms: 1: active intervention
Drug: Indomethacin — 25, 50 or 75 mg, PO. Singe dose.
  Other Names: Indocin
  Arms: 1: active intervention
Drug: Ibuprofen — 300, 600 or 900 mg, PO. Single dose.
  Other Names: Advil, Motrin
  Arms: 1: active intervention
Drug: Oxymetazoline 0.05% nasal solution — 1-2 sprays/ nostril. Single dose.
  Other Names: Afrin
  Arms: 1: active intervention
Dietary Supplement: Bovril — 6-10 g, PO. Single dose.
  Arms: 1: active intervention
Drug: Acetazolamide — 125-1000 mg PO. Single dose. Alone or in combination with yohimbine or midodrine
  Other Names: Diamox
  Arms: 1: active intervention
Drug: Rivastigmine tartrate — 1.5-6 mg PO. Single dose.
  Other Names: Exelon
  Arms: 1: active intervention
Drug: Carbidopa/levodopa — 10mg/100mg or 25mg/100mg. 1-2 tab PO. Single dose. Alone or in combination with carbidopa (Lodosyn) 25-175 mg
  Other Names: Sinemet, Lodosyn
  Arms: 1: active intervention
Device: Inflatable abdominal binder — External abdominal compression (20-40 mm Hg) with an inflatable abdominal binder applied after a pressor agent (e.g. midodrine, yohimbine).
  Other Names: external abdominal compression
  Arms: 1: active intervention
Device: inflatable abdominal binder (sham) — External abdominal compression (5 mm Hg) with an inflatable abdominal binder applied after a pressor agent (e.g. midodrine, yohimbine).
  Other Names: external abdominal compression (sham)
  Arms: 2: Placebo or sham device

SUMMARY:
The autonomic nervous system serves multiple regulatory functions in the body, including the regulation of blood pressure and heart rate, gut motility, sweating and sexual function. There are several diseases characterized by abnormal function of the autonomic nervous system. Medications can also alter autonomic function. Impairment of the autonomic nervous system by diseases or drugs may lead to several symptoms, including blood pressure problems (e.g., high blood pressure lying down and low blood pressure on standing), sweating abnormalities, constipation or diarrhea and sexual dysfunction. Because treatment options for these patients are limited. We propose to study patients autonomic failure and low blood pressure upon standing and determine the cause of their disease by history and examination and their response to autonomic testing which have already been standardized in our laboratory. Based on their possible cause, we will tests different medications that may alleviate their symptoms.

DETAILED DESCRIPTION:
Subjects will be admitted to the Clinical Research Center at Vanderbilt University for the studies. The average inpatient stay is 7 days. Initially a complete history and physical will be performed and the patient will be placed on a low monamine, no methylxanthine, 150 mEq sodium, 60-80 mEq potassium diet.

The following tests will be performed:

1. Meal challenge:

   We observed profound effects of diet on blood pressure in many patients with orthostatic hypotension. Some patients dropped their blood pressure by 40-60 mmHg during the postprandial period. Blood pressure will be monitored with an automated device (Dinamap) after feeding the patients with a standardized diet.
2. Physiologic autonomic tests:

   Patients are studied supine, and blood pressure is monitored with a sphygmomanometer or an automated device (Dinamap, Finapres or tonometer).
   1. Orthostatic test: Blood pressure and heart rate are measured in the supine and standing positions. Orthostatic hypotension without an adequate heart rate increase is indicative of autonomic failure. On the other hand, orthostatic tachycardia in the absence of volume depletion is seen in "hyperadrenergic orthostatic hypotension".
   2. Standing time: The time the patient can stand motionless gives a very good indication of functional capacity.
   3. Deep breathing: Heart rate is monitored with an ECG and the patient is asked to breathe deeply 6 times each minute for two minutes. Heart rate variation due to respiration is an autonomic function. The loss of this respiratory arrhythmia is indicative of autonomic failure.
   4. Valsalva maneuver: The patient is asked to exhale against a 40 mmHg pressure. This produces transient changes in blood pressure and heart rate which are autonomically mediated, and can be monitored with an ECG. Failure to observe heart rate changes is indicative of autonomic failure.
   5. Hyperventilation: The patient is asked to hyperventilate for 30 seconds. The normal response is an increase in heart rate and no significant change in blood pressure. Patients with autonomic failure have profound reductions in blood pressure without compensatory heart rate increases.
   6. Handgrip: The patient is asked to maintain a handgrip for three minutes. Increases in heart rate and blood pressure are seen in normal subjects but not in patients with autonomic failure.
   7. Cold pressor test: The patient is asked to place an hand in ice cold water for one minute. The results are similar to the handgrip test.
   8. Supine hypertension screening: We will measure the blood pressure every two hours during one night to determine if the patient has supine hypertension or high blood pressure while lying down.
3. Posture Study:

   Blood for catecholamine, bradykinins, plasma renin activity, aldosterone and plasma angiotensin II is drawn while the patient is supine and upright. Blood pressure is measured with a sphygmomanometer or an automated device (Dinamap). Normally, on assuming the upright posture, plasma norepinephrine and renin activity should double. Patients with autonomic failure typically show low supine levels of both norepinephrine and renin activity which failed to increase on assuming the upright posture. In contrast, patients with hyperadrenergic orthostatic hypotension typically have normal or exaggerated responses.
4. Twelve hour urine collections for catecholamines, urinalysis, protein, glucose, creatinine, osmolality, electrolytes and F2-isoprostanes will be collected to analyze for catecholamine excretion (hormones produces by the autonomic nervous system) oxidative stress markers and to assess the patient's kidney function.
5. Blood will be collected in the fasted state through and intravenous catheter to analyze for PAI-1, CRP, F2-isoprostanes, proinflammatory cytokines and renal function.
6. EKG will be recorded while the patient is lying down and while the patient is standing.
7. Orthostatic vital signs will be measured several times a day. This testing consists of blood pressure and heart rate measured while the patient is lying down and then repeated after standing quietly for 10 minutes. Several readings are measured in sequence using an automated blood pressure monitor (Dinamap).
8. Tilt table test: This test uses a tilt table, which is a motorized table with a footboard. The participant rests quietly on the table while the monitoring equipment is assembled. EKG electrodes are applied to the chest to monitor heart rate and rhythm. Blood pressure will be measured with a cuff applied to a finger. Blood pressure will also be checked periodically using a traditional blood pressure cuff wrapped around an upper arm. Safety straps are used to secure the patient to the table to prevent falling or unsteadiness when the table is moved to an upright position. Gradual head up tilt will be performed until a systolic blood pressure of 70 mm Hg is reached or the appearance of symptoms related to hypotension. Changes in cardiac output (heart's pumping capacity) will be measured by analyzing the air that is breathed ("rebreathing test", Innocor). This will be done through a mouthpiece connected to a bag full of air and small concentrations of the inactive gases SF6 and N2O. Subjects will breathe normally through a mouthpiece connected to a bag for about 5 minutes at baseline, at 30º and at the maximum head up tilt. Innocor is FDA approved for inert gases cardiac output measurement.

   This test may or may not be performed. Some patients may have already undergone this test or it may not be pertinent to a particular patient. The principal investigator will decide whether this test is performed or not.
9. Therapeutic Drug Trials:

We will try different medications to determine if blood pressure improves upon standing. For all these tests, blood pressure is monitored with a sphygmomanometer and heart rate with an ECG. The procedures are detailed below.

Patients will be in the fasted state in the seated position throughout the study. They will be connected to an automated blood pressure monitor (Dinamap). Thirty minutes after baseline blood pressure and heart rate measurements, they will be given a dose of the medicine to be tested. Blood pressure will be monitored every 5 to 15 minutes for up to four additional hours. Upright blood pressure, heart rate and the standing time will be measure periodically throughout the study. The patients will be asked to rate their symptoms at various time during the study.

This study has been designed to determine optimal candidate drugs and therapy for the treatment of orthostatic hypotension. Potential pressor agents have been selected for this study because of their different mechanism of action. We propose also to use the combination of different therapeutic agents.

For some of these tests,we will do the following:

1. we will determine the effect of the medication on catecholamines and/or markers of inflammation and/or oxidative stress. We will draw a blood sample at baseline and after the medication has taken effect. A saline lock or small flexible intravenous catheter will be placed for this purpose. For each medication trial, the amount of blood drawn would be up to 6 teaspoons. The total blood drawn for all the medication trials would not exceed 36 teaspoons.
2. We will apply external abdominal compression (up to 40mm Hg) to evaluate the ability of this counterpressure method in combination with a pressor agent to improve orthostatic tolerance. For this purpose, we will use an abdominal binder with an inflatable cuff placed underneath, which will be inflated to exert pressure at the level of the umbilicus while patients are standing. Patients may be randomly assigned to 5mm Hg (sham treatment) and/or 20-40mm Hg external abdominal compression with an abdominal binder applied at baseline of some of the therapeutic trials described above. The principal investigator will decide which medication will be used in each trial.
3. We will measure changes in cardiac output (heart's pumping capacity) by analyzing the air that is breathed ("rebreathing test", Innocor). This will be done through a mouthpiece connected to a bag full of air and small concentrations of the inactive gases SF6 and N2O. Subjects will breathe normally through a mouthpiece connected to a bag for about 5 minutes before and after the medication. Innocor is FDA approved for inert gases cardiac output measurement.
4. We will measure the cerebral blood flow to determine if it can be improved with the medication. A middle cerebral artery will be continuously insonated by transcranial Doppler ultrasonography. The transducer will be affixed with head straps.
5. We will apply eleven sticky patches to the front of the body to measure the impedance (electrical resistance). This will allow us to determine fluid shifts between body segments and obtain a continuous measurement of cardiac output and peripheral resistance.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for evaluation of their autonomic function
* Ages 18-85

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2002-03; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Increase in seated systolic blood pressure 1-hr post drug compared to baseline. | 1.5-4 hours

SECONDARY OUTCOMES:
Increase in standing time 1-hr post drug compared to baseline | 1.5-4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Background] Shibao C, Okamoto L, Biaggioni I. Pharmacotherapy of autonomic failure. Pharmacol Ther. 2012 Jun;134(3):279-86. doi: 10.1016/j.pharmthera.2011.05.009. Epub 2011 Jun 12. PMID 21664375
- [Background] Garland EM, Hooper WB, Robertson D. Pure autonomic failure. Handb Clin Neurol. 2013;117:243-57. doi: 10.1016/B978-0-444-53491-0.00020-1. PMID 24095130
- [Background] Arnold AC, Biaggioni I. Management approaches to hypertension in autonomic failure. Curr Opin Nephrol Hypertens. 2012 Sep;21(5):481-5. doi: 10.1097/MNH.0b013e328356c52f. PMID 22801444
- [Result] Jordan J, Shannon JR, Biaggioni I, Norman R, Black BK, Robertson D. Contrasting actions of pressor agents in severe autonomic failure. Am J Med. 1998 Aug;105(2):116-24. doi: 10.1016/s0002-9343(98)00193-4. PMID 9727818
- [Result] Shibao C, Gamboa A, Diedrich A, Biaggioni I. Management of hypertension in the setting of autonomic failure: a pathophysiological approach. Hypertension. 2005 Apr;45(4):469-76. doi: 10.1161/01.HYP.0000158835.94916.0c. Epub 2005 Feb 28. PMID 15738343
- [Result] Shibao C, Arzubiaga C, Roberts LJ 2nd, Raj S, Black B, Harris P, Biaggioni I. Hyperadrenergic postural tachycardia syndrome in mast cell activation disorders. Hypertension. 2005 Mar;45(3):385-90. doi: 10.1161/01.HYP.0000158259.68614.40. Epub 2005 Feb 14. PMID 15710782
- [Result] Jordan J, Shannon JR, Diedrich A, Black B, Robertson D, Biaggioni I. Water potentiates the pressor effect of ephedra alkaloids. Circulation. 2004 Apr 20;109(15):1823-5. doi: 10.1161/01.CIR.0000126283.99195.37. Epub 2004 Apr 5. PMID 15066944
- [Result] Jacob G, Costa F, Biaggioni I. Spectrum of autonomic cardiovascular neuropathy in diabetes. Diabetes Care. 2003 Jul;26(7):2174-80. doi: 10.2337/diacare.26.7.2174. PMID 12832331
- [Result] Biaggioni I, Robertson RM. Hypertension in orthostatic hypotension and autonomic dysfunction. Cardiol Clin. 2002 May;20(2):291-301, vii. doi: 10.1016/s0733-8651(01)00005-4. PMID 12119802
- [Result] Jordan J, Biaggioni I. Diagnosis and treatment of supine hypertension in autonomic failure patients with orthostatic hypotension. J Clin Hypertens (Greenwich). 2002 Mar-Apr;4(2):139-45. doi: 10.1111/j.1524-6175.2001.00516.x. PMID 11927799
- [Result] Shannon JR, Diedrich A, Biaggioni I, Tank J, Robertson RM, Robertson D, Jordan J. Water drinking as a treatment for orthostatic syndromes. Am J Med. 2002 Apr 1;112(5):355-60. doi: 10.1016/s0002-9343(02)01025-2. PMID 11904109
- [Result] Jordan J, Shannon JR, Black BK, Ali Y, Farley M, Costa F, Diedrich A, Robertson RM, Biaggioni I, Robertson D. The pressor response to water drinking in humans : a sympathetic reflex? Circulation. 2000 Feb 8;101(5):504-9. doi: 10.1161/01.cir.101.5.504. PMID 10662747
- [Result] Shibao C, Gamboa A, Diedrich A, Dossett C, Choi L, Farley G, Biaggioni I. Acarbose, an alpha-glucosidase inhibitor, attenuates postprandial hypotension in autonomic failure. Hypertension. 2007 Jul;50(1):54-61. doi: 10.1161/HYPERTENSIONAHA.107.091355. Epub 2007 May 21. PMID 17515447
- [Result] Shibao C, Raj SR, Gamboa A, Diedrich A, Choi L, Black BK, Robertson D, Biaggioni I. Norepinephrine transporter blockade with atomoxetine induces hypertension in patients with impaired autonomic function. Hypertension. 2007 Jul;50(1):47-53. doi: 10.1161/HYPERTENSIONAHA.107.089961. Epub 2007 May 21. PMID 17515448
- [Result] Shibao C, Okamoto LE, Gamboa A, Yu C, Diedrich A, Raj SR, Robertson D, Biaggioni I. Comparative efficacy of yohimbine against pyridostigmine for the treatment of orthostatic hypotension in autonomic failure. Hypertension. 2010 Nov;56(5):847-51. doi: 10.1161/HYPERTENSIONAHA.110.154898. Epub 2010 Sep 13. PMID 20837887
- [Result] Okamoto LE, Shibao C, Gamboa A, Choi L, Diedrich A, Raj SR, Black BK, Robertson D, Biaggioni I. Synergistic effect of norepinephrine transporter blockade and alpha-2 antagonism on blood pressure in autonomic failure. Hypertension. 2012 Mar;59(3):650-6. doi: 10.1161/HYPERTENSIONAHA.111.184812. Epub 2012 Feb 6. PMID 22311903
- [Derived] Okamoto LE, Walsh E, Diedrich A, Shibao CA, Gamboa A, Black BK, Paranjape SY, Muldowney JA 3rd, Habermann R, Peltier A, Tarpara K, Biaggioni I. Clinical Correlates of Efficacy of Pyridostigmine in the Treatment of Orthostatic Hypotension. Hypertension. 2025 Mar;82(3):489-497. doi: 10.1161/HYPERTENSIONAHA.124.24050. Epub 2024 Dec 27. PMID 39727053
- [Derived] Okamoto LE, Diedrich A, Baudenbacher FJ, Harder R, Whitfield JS, Iqbal F, Gamboa A, Shibao CA, Black BK, Raj SR, Robertson D, Biaggioni I. Efficacy of Servo-Controlled Splanchnic Venous Compression in the Treatment of Orthostatic Hypotension: A Randomized Comparison With Midodrine. Hypertension. 2016 Aug;68(2):418-26. doi: 10.1161/HYPERTENSIONAHA.116.07199. Epub 2016 Jun 6. PMID 27271310